CLINICAL TRIAL: NCT02550106
Title: A Phase IV, Multicenter, Single-arm and Open-label Study With Omalizumab (Xolair®) in Chronic Spontaneous Urticaria (CSU) Patients Who Remain Symptomatic Despite Antihistamine (H1) Treatment
Brief Title: Omalizumab in Chronic Spontaneous Urticaria Patients Non Responding to Initial Standard antihistaminE Treatment
Acronym: SUNRISE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CIGE025EFR02
Record Dates: First submitted 2015-03-09; First posted 2015-09-15 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: CHRONIC SPONTANEOUS URTICARIA
Keywords: CHRONIC SPONTANEOUS URTICARIA; OMALIZUMAB; URTICARIA CONTROL TEST; IGE025
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OMALIZUMAB (Experimental): sub cutaneous injections of 300 mg every 4 weeks until Week 8.
  Interventions: Drug: OMALIZUMAB

INTERVENTIONS:
Drug: OMALIZUMAB — sub cutaneous injections of 300 mg every 4 weeks until Week 8.

SUMMARY:
Evaluate the proportion of patients with an urticaria control test [UCT] score of greater than or equal to 12 at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 75 years.
* Diagnosis of CSU for ≥ 6 months and an inadequate response to nsH1 antihistamines at the time of the request, as defined by the following:
* The presence of itch and hives for > 6 consecutive weeks at any time prior to enrollment, despite current use of H1 antihistamine therapy during this time period.
* Weekly UAS7 score (range 0 to 42) 16 and UCT score (range 0 to 16) < 8 prior to enrollment (Day 1)
* Current use of an H1 antihistamine for CSU on the day of the initial visit and Day
* Informed consent

Exclusion Criteria:

* Treatment with an investigational agent within 30 days before enrollment.
* Routine (daily or every other day during 5 or more consecutive days) doses of the following medications within 30 days prior to Day -7: systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide.
* Intravenous (i.v.) immunoglobulin G or plasmapheresis within 30 days prior to Day -7
* Regular (daily/every other day) doxepin (oral) use within 14 days prior to Day -7.
* Any H2 antihistamine use within 7 days prior to Day -7.
* Any leukotriene receptor antagonist (LTRA) (montelukast or zafirlukast) within 7 days prior to Day 7.
* Concomitant use of cyclosporine or any other immunosuppressive agent.
* Hypersensitivity to omalizumab or any component of the formulation.
* History of anaphylactic shock.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2015-04-22 (Actual); Primary Completion 2016-01-11 (Actual); Study Completion 2016-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CLAIRE BERNIER TAUGOURDEAU, Principal Investigator — HOPITAL HOTEL DIEU - NANTES CEDEX 1; PASCAL JOLY, Principal Investigator — HOPITAL CHARLES NICOLLE - ROUEN CEDEX; LUDOVIC MARTIN, Principal Investigator — HOTEL DIEU - ANGERS CEDEX 9; GERARD GUILLET, Principal Investigator — CHR LA MILETRIE - POITIERS CEDEX; PATRICE PLANTIN, Principal Investigator — CHI DE CORNOUAILLE - QUIMPER CEDEX; ALAIN DUPUY, Principal Investigator — HOPITAL PONTCHAILLOU - RENNES CEDEX 9; EVELYNE COLLET, Principal Investigator — CHU SITE DU BOCAGE - DIJON CEDEX; ANNICK BARBAUD, Principal Investigator — HOPITAUX DE BRABOIS - VANDOEUVRE LES NANCY CEDEX; ZIAD REGUIAI, Principal Investigator — HOPITAL ROBERT DEBRE - REIMS CEDEX; FABIEN PELLETIER, Principal Investigator — HOPITAL JEAN MINJOZ - BESANCON CEDEX; DELPHINE STAUMONT SALLE, Principal Investigator — HOPITAL CLAUDE HURIEZ- LILLE CEDEX; JULIETTE JEGOU, Principal Investigator — CH DE CHALONS EN CHAMPAGNE - CHALONS EN CHAMPAGNE CEDEX; EMMANUELLE AMSLER, Principal Investigator — HOPITAL TENON - PARIS CEDEX 20; OLIVIER CHOSIDOW, Principal Investigator — HOPITAL HENRI MONDOR - CRETEIL; VINCENT DESCAMPS, Principal Investigator — HOPITAL BICHAT CLAUDE BERNARD - PARIS CEDEX 18; EMMANUEL MAHE, Principal Investigator — CH VICTOR DUPOUY - ARGENTEUIL CEDEX; LILIANE LAROCHE, Principal Investigator — HOPITAL AVICENNE - BOBIGNY CEDEX; GERMAINE GABISON, Principal Investigator — HOPITAL SAINT LOUIS - PARIS CEDEX 10; SELIM ARACTINGI, Principal Investigator — HOPITAL COCHIN - PARIS; LAURENCE BOUILLET, Principal Investigator — CHU DE GRENOBLE - LA TRONCHE; JEAN-JACQUES GROB, Principal Investigator — HOPITAL TIMONE - MARSEILLE CEDEX 05; FREDERIC CAMBAZARD, Principal Investigator — CHU SAINT ETIENNE - ST PRIEST EN JAREZ CEDEX; THIERRY BOYE, Principal Investigator — HIA SAINTE ANNE - TOULON CEDEX 9; JEAN-PHILIPPE LACOUR, Principal Investigator — HOPITAL DE L'ARCHET - NICE CEDEX 3; PHILIPPE BERBIS, Principal Investigator — HOPITAL NORD- MARSEILLE; LAURENT MEUNIER, Principal Investigator — HOPITAL CAREMEAU - NIMES CEDEX 9; FRANCOISE GIORDANO LABADIE, Principal Investigator — HOPITAL LARREY - TOULOUSE CEDEX 9; NADIA RAISON PEYRON, Principal Investigator — HOPITAL ST ELOI - MONTPELLIER CEDEX 5; MARIE CHRISTINE FERRIER LE BOUEDEC, Principal Investigator — CHU ESTAING - CLERMONT FERRAND; MARIE SYLVIE DOUTRE, Principal Investigator — HOPITAL DE HAUT LEVEQUE - PESSAC CEDEX; BRIGITTE MILPIED, Principal Investigator — HOPITAL ST ANDRE - BORDEAUX CEDEX; CHRISTOPHE BEDANE, Principal Investigator — HOPITAL DUPUYTREN - LIMOGES CEDEX 1; PHILIPPE MODIANO, Principal Investigator — HOPITAL ST VINCENT DE PAUL - LILLE CEDEX
Locations (27):
- France (27):
  - Novartis Investigative Site, Paris, Cedex 10
  - Novartis Investigative Site, Limoges, Haute Vienne
  - Novartis Investigative Site, Toulon, Val De Marne
  - Novartis Investigative Site, Angers
  - Novartis Investigative Site, Argenteuil
  - Novartis Investigative Site, Besançon
  - Novartis Investigative Site, Bobigny
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Châlons-en-Champagne
  - Novartis Investigative Site, Clermont-Ferrand
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Nîmes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Quimper
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Rouen
  - Novartis Investigative Site, Saint-Etienne
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Vandœuvre-lès-Nancy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Full Analysis Set
Period: Overall Study
Arm/Group | OMALIZUMAB
Started | 136
Completed | 124
Not Completed | 12
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 3
Not completed — Protocol Violation | 6
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | OMALIZUMAB
Number analyzed (Participants) | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106
  Male | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With an Urticaria Control Test [UCT] Score of Greater Than or Equal to 12
Description: Number of participants with an Urticaria Control Test score of greater than or equal to 12 at Week 12
  The UCT is a simple 4-item tool. A score between 0 and 4 is assigned to every answer option. Subsequently, the scores for all 4 questions are summed up. Accordingly, the minimum and maximum UCT scores are 0 and 16, with 16 points indicating complete disease control.
Time Frame: WEEK 12
Population: (Full analysis set, LOCF)
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- OMALIZUMAB With ANGIOEDEMA: sub cutaneous injections of 300 mg every 4 weeks until W8
Arm/Group | OMALIZUMAB With ANGIOEDEMA
Number analyzed (Participants) | 136
percent of participants | 75.0 [66.9 to 82.0]

2. Secondary Outcome: Percent of Participants With UAS7≤6 (Patients Achieving Disease Control), in Adult Patients With CSU, With or Without the Presence of Angioedema
Description: 2 patients with angioedema status were missing at baseline and not included
Time Frame: WEEK 12
Population: Full Analysis Set
  2 patients with angioedema status missing at baseline were not included so that FAS = 83 + 51 + 2= 136
Measure: Number (95% Confidence Interval); unit: percent of participants
Groups:
- OMALIZUMAB Without Angioedema: sub cutaneaous injections of 300 mg every 4 weeks until Week 8
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without Angioedema
Number analyzed (Participants) | 83 | 51
percent of participants | 69.6 [58.2 to 79.5] | 63.8 [48.5 to 77.3]

3. Secondary Outcome: CSU Disease Activity Using the Urticaria Activity Score (UAS7), With or Without the Presence of Angioedema
Description: A total score of UAS7 is calculated by adding for 7 days the daily UAS. The UAS7 is the sum of the daily UAS over 7 days before baseline and W12. The UAS7 score ranges from 0 to 42 with higher scores reflecting higher activity of the disease.
  Scores were categorized into five diseases states : urticaria-free (score =0), well-controlled (scores 1-6), mild (scores 7-15), moderate (scores 16-27) and severe urticaria (scores 28-42).
Time Frame: baseline and week 12
Population: Full Analysis Set (FAS)
Measure: Mean (Standard Deviation); unit: scores on a scale
Groups:
- OMALIZUMAB Without ANGIOEDEMA: sub cutaneous injections of 300 mg every 4 weeks until W8
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 79 | 47
scores on a scale
  baseline | 29.7 (7.32) | 29.2 (6.72)
  at week 12 | 6.6 (10.08) | 6.5 (9.11)

4. Secondary Outcome: Urticaria Control Test (UCT) Score According to the Presence of Angioedema at Baseline and Week 12
Description: The UCT is a questionnaire collecting retrospective information over the last 4 weeks before baseline and W12.
  The UCT score ranges from 0 to 16 with higher scores reflecting lower control of the disease.
  A score of ≥12 indicates well-controlled urticaria.
Time Frame: baseline and week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 82 | 50
scores on a scale
  baseline | 3.0 (2.06) | 3.6 (2.55)
  at week 12 | 13.1 (3.95) | 12.9 (3.97)

5. Secondary Outcome: Control of the CSU Using the UCT Score for Patients in Extension Treatment Period Phase at Week 16, With or Without the Presence of Angioedema
Description: The UCT is a simple 4-item tool. A score between 0 and 4 is assigned to every answer option. Subsequently, the scores for all 4 questions are summed up. Accordingly, the minimum and maximum UCT scores are 0 and 16, with 16 points indicating complete disease control.
Time Frame: week 16
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 70 | 42
scores on a scale | 14.2 (2.96) | 13.4 (3.40)

6. Secondary Outcome: Control of the CSU Using the UCT Score for Patients in Extension Treatment Period Phase at Week 20, With or Without the Presence of Angioedema
Description: as for outcome 5
Time Frame: week 20
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 48 | 34
scores on a scale | 14.4 (2.40) | 13.3 (4.11)

7. Secondary Outcome: Control of the CSU Using the UCT Score for Patients in Extension Treatment Period Phase at Week 24, With or Without the Presence of Angioedema
Description: as for outcome 5
Time Frame: week 24
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 14 | 12
scores on a scale | 14.5 (2.14) | 13.4 (3.75)

8. Secondary Outcome: Control of the CSU Using the UCT Score for Patients in Extension Treatment Period Phase at Week 28, With or Without the Presence of Angioedema
Description: as for outcome 5
Time Frame: week 28
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 2 | 2
scores on a scale | 13.5 (3.54) | 12.0 (5.66)

9. Secondary Outcome: The Quality of Life Using the Chronic Urticaria Quality of Life (CU-QoL) Questionnaire
Description: The Cu-QoL is a questionnaire collecting retrospective information over the last 2 weeks before baseline and W12.
  The CU-QoL total score is transformed to range from 0 to 100, with higher scores indicating worse Health Related Quality of life.
Time Frame: baseline and week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without ANGIOEDEMA
Number analyzed (Participants) | 80 | 49
scores on a scale
  baseline | 68.9 (15.64) | 62.4 (17.76)
  at 12 weeks | 32.5 (13.33) | 33.3 (13.32)

10. Secondary Outcome: The Angioedema Quality of Life (AE-QoL)
Description: The angioedema Quality of Life Questionnaire is a valuable tool to assess changes of QoL impairment in angioedema patients.
  The results of all the answered questions are summed up and transferred to a scale ranging from 0 to 100, with higher scores indicative of a higher QoL impairment
Time Frame: baseline and week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA
Number analyzed (Participants) | 78
scores on a scale
  baseline | 57.88 (22.474)
  at week 12 | 16.40 (20.074)

11. Secondary Outcome: The Dermatology Life Quality Index (DLQI)
Description: The Dermatology life Quality Index (DLQI) is a ten-question questionnaire used to measure the impact of skin disease on the quality of life of an affected person. It is designed for people aged 16 years and above. Each question is scored from 0 to 3, giving a possible score range form 0 (meaning no impact of skin disease on quality of life) to 30 (meaning maximum impact on quality of life).
Time Frame: baseline and week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA | OMALIZUMAB Without Angioedema
Number analyzed (Participants) | 79 | 49
scores on a scale
  baseline | 14.2 (5.39) | 13.2 (6.67)
  at week 12 | 2.4 (3.95) | 2.7 (5.12)

12. Secondary Outcome: Angioedema Activity Using the Angioedema Activity Score (AAS)
Description: The Angioedema Activity Score (AAS) was completed by patients on a daily basis. The AAS is a validated questionnaire to determine the severity and impact of the angioedema episode. Te daily AAS values are added over 7 days before baseline and W12. Weekly AAS (AAS7) scores range from 0 to 105, with higher scores indicative of a higher disease activity.
Time Frame: baseline and week 12
Population: FAS
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | OMALIZUMAB With ANGIOEDEMA
Number analyzed (Participants) | 78
scores on a scale
  baseline | 32.7 (27.21)
  at week 12 | 3.7 (10.40)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment at week 12
Description: An adverse event (AE) is any sign or symptom that occurs during the study treatment plus the # days post treatment
Groups:
- Omalizumab 300 mg: Omalizumab 300 mg
Arm/Group | Omalizumab 300 mg
Serious Adverse Events (participants affected / at risk) | 9/136
Other Adverse Events (participants affected / at risk) | 44/136
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 300 mg (N=136)
PNEUMONIA (Infections and infestations) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
FRACTURED SACRUM (Injury, poisoning and procedural complications) | 1
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1
OBESITY (Metabolism and nutrition disorders) | 1
FOOT DEFORMITY (Musculoskeletal and connective tissue disorders) | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1
SACROILIITIS (Musculoskeletal and connective tissue disorders) | 1
BLADDER DILATATION (Renal and urinary disorders) | 1
URINARY INCONTINENCE (Renal and urinary disorders) | 1
PHARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omalizumab 300 mg (N=136)
ASTHENIA (General disorders) | 23
WEIGHT INCREASED (Investigations) | 7
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 12
HEADACHE (Nervous system disorders) | 22

LIMITATIONS AND CAVEATS:
No placebo arm and limited duration of the study (3 months for the main period)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial